CLINICAL TRIAL: NCT07040410
Title: The Effect of Aromatherapy and Music on Pain, Vital Signs and Parental Satisfaction in Children Undergoing Peritoneal Dialysis Treatment: A Randomized Controlled Study
Brief Title: Aromatherapy and Music on Pain, Vital Signs and Parental Satisfaction in Children Undergoing Peritoneal Dialysis
Acronym: 2024-KAEK-11
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Eda Aktaş, PhD, RN, Associate Professor, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: KAEK-11/30.04.2025.142; KAEK-11/30.04.2025.142 (Other: Başakşehir Çam and Sakura City Hospital)
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Pain; Vital Signs Monitoring; Parental Satisfaction
Keywords: peritoneal dialysis treatment; pain management; pain in children; non-pharmacological method; satisfaction
MeSH Terms: conditions — Pain; Agnosia; Personal Satisfaction | interventions — Aromatherapy; Music Therapy

STUDY DESIGN:
Intervention Model Description: This study is designed as an interventional, cross-over, randomized-controlled design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aromatherapy (Experimental): Fifteen minutes before the PD session and during the first outflow and inflow phases, aromatherapy will be administered via inhalation. Five drops of 100% pure organic lavender oil will be added to drinking water in a diffuser visible to the child and parent. The diffuser will be plugged in at the bedside, and participants will be warned not to touch the device. Pain and vital signs will be assessed as in the control group.
  Interventions: Procedure: Aromatherapy
- Music Therapy (Experimental): Fifteen minutes before the PD session and during the first outflow and inflow phases, music chosen by the child or parent will be played. Pain and vital signs will be assessed as in the control group.
  Interventions: Procedure: Music Therapy
- Control (Experimental): Peritoneal dialysis treatment will be started with discharge first, and then the amount of dialysate fluid determined by the physician's request will be filled. In the clinical routine, nonpharmacological pain treatment method is not applied during excretion and filling. Nonpharmacological pain treatment method will not be applied to the control group. The "Wong-Baker Facial Expressions Rating Scale" and "Life Signs Evaluation Form" will be filled in by the researcher at the 0th and 1st minutes of the first discharge and at the 0th and 1st minutes of the first filling.
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Aromatherapy — Fifteen minutes before the PD session and during the first outflow and inflow phases, aromatherapy will be administered via inhalation. Five drops of 100% pure organic lavender oil
  Arms: Aromatherapy
Procedure: Music Therapy — Fifteen minutes before the PD session and during the first outflow and inflow phases, music chosen by the child or parent will be played. Pain and vital signs will be assessed as in the control group.
  Arms: Music Therapy
Procedure: Control — Peritoneal dialysis treatment will be started with discharge first, and then the amount of dialysate fluid determined by the physician's request will be filled. In the clinical routine, nonpharmacological pain treatment method is not applied during excretion and filling. Nonpharmacological pain treatment method will not be applied to the control group. The "Wong-Baker Facial Expressions Rating Scale" and "Life Signs Evaluation Form" will be filled in by the researcher at the 0th and 1st minutes of the first discharge and at the 0th and 1st minutes of the first filling.
  Arms: Control

SUMMARY:
This study is an experimental randomized controlled study conducted to compare the effect of two different nonpharmacological treatment methods (aromatherapy and music therapy) on pain, vital signs and parental satisfaction to alleviate or eliminate pain during excretion and filling in children undergoing peritoneal dialysis treatment. The study population consists of pediatric patients aged 3 to 18 years undergoing peritoneal dialysis treatment at Basaksehir Cam and Sakura City Hospital between June 2025- 2026. According to literature, for experimental studies and parametric measurements, at least 30 participants should be included in both experimental and control groups. Therefore, this crossover randomized design will include 45 children per group: control, aromatherapy, and music therapy. Children included in the sample will be assigned to groups based on a crossover randomized design. This method is suitable for studies with a small sample size. Since three different interventions will be applied once per session over three sessions, to avoid bias, the order of interventions will be randomized and labeled as A, B, and C. The researcher will write the names of the interventions on three separate papers, draw them one by one, and assign them accordingly: Method A: Aromatherapy, Method B: Music Therapy, Method C: Control. Then, the six possible sequences (ABC, ACB, BAC, BCA, CAB, CBA) will be written on six papers and drawn randomly to determine the intervention order for each participant.

DETAILED DESCRIPTION:
The study is a randomized controlled, non-blinded, experimental trial. The study population consists of pediatric patients aged 3 to 18 years undergoing peritoneal dialysis treatment at Basaksehir Cam and Sakura City Hospital between June 2025-2026. According to literature, for experimental studies and parametric measurements, at least 30 participants should be included in both experimental and control groups. Therefore, this crossover randomized design will include 45 children per group: control, aromatherapy, and music therapy. Children included in the sample will be assigned to groups based on a crossover randomized design. In order to prevent bias and increase the validity of the data, the pain scores of the children before and after the procedure were assessed by three different groups as children participating in the study (n:45), their parents as the people who know the children best (n:45), and a researcher specialized in pediatric nursing (n:1), and the inter-observer agreement was examined.

The data collection phase of the research is planned to be completed between June 2025-2026.In this experimental study, the children and their parents who came to the nephrology clinics were evaluated in terms of the inclusion criteria and the children and parents who did not meet the criteria were excluded from the study. The children and parents complying with the inclusion criteria were informed about the study and their written and verbal consents were received. Pre-application will be made before starting the data collection process.

Pilot Study Phase: Children and parents meeting the inclusion criteria will be informed about the study and their verbal and written consent will be obtained. A pilot will be conducted with five children. Based on the results, data collection tools will be revised if necessary.

Pre-Implementation Phase: Children and parents included in the sample will be informed about the study. Written and verbal consent will be obtained. The "Descriptive Information Form" and "Vital Signs Evaluation Form" will be completed by the researcher before the peritoneal dialysis session begins. To avoid causing additional pain, no invasive procedure will be performed within 30 minutes prior to the PD session. Group assignments will be determined through randomization. The PD session will be performed in accordance with physician recommendations.

Implementation Phase: To eliminate variation from different nursing techniques, data collection and application of non-pharmacological interventions will be carried out solely by the researcher. Each child will participate in the control, aromatherapy, and music therapy groups in a randomized order (n = 45 per group).

Control Group: Peritoneal dialysis treatment will be started with discharge first, and then the amount of dialysate fluid determined by the physician's request will be filled. In the clinical routine, nonpharmacological pain treatment method is not applied during excretion and filling. Nonpharmacological pain treatment method will not be applied to the control group. The "Wong-Baker Facial Expressions Rating Scale" and "Life Signs Evaluation Form" will be filled in by the researcher at the 0th and 1st minutes of the first discharge and at the 0th and 1st minutes of the first filling.

Aromatherapy Group: Fifteen minutes before the PD session and during the first outflow and inflow phases, aromatherapy will be administered via inhalation. Five drops of 100% pure organic lavender oil will be added to drinking water in a diffuser visible to the child and parent. The diffuser will be plugged in at the bedside, and participants will be warned not to touch the device. Pain and vital signs will be assessed as in the control group.

Music Therapy Group: Fifteen minutes before the PD session and during the first outflow and inflow phases, music chosen by the child or parent will be played. Pain and vital signs will be assessed as in the control group.

Post-Implementation Phase: After completing the assigned intervention and while the dialysate dwells in the peritoneum, no additional non-pharmacological methods will be applied. During this phase, the Parental Satisfaction Questionnaire will be completed by the researcher. Data collection will conclude once the required sample size is reached. The study followed the CONSORT guideline for reporting randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Children will be included between the ages of 3 and 18 who receive instrumental peritoneal dialysis or continuous outpatient peritoneal dialysis treatment.
* Children who have a sufficient cognitive level (3-18 years) to determine pain scores,
* Children who have a healthy hearing and vision system,
* Children who did not take painkillers, opioids or sedatives 6 hours before the study,
* Children who have absence of severe pain in another part of the body,
* Children who have absence of a history of allergies,
* Children and parents who can speak and understand Turkish.

Exclusion Criteria:

* Decline to participate in the study,
* Peritonitis diagnosis,
* Pain due to catheter immobilization,
* Receiving the first session of peritoneal dialysis treatment

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Pain severity | 12 months
  The children and the parents were informed about the Wong Baker Faces Pain Rating Scale and they were asked to mark the children's pain levels on the scale. In addition, the pain levels of the children before and after the procedure were determined by the researcher who is a specialist in pediatric nursing by using the same scales. The scale will be applied at 0 and 1 minute of the first outflow and inflow phases by the researcher.

SECONDARY OUTCOMES:
Heart Rate Monitoring | 12 months
  Developed by the researchers, this form records heart rate using a Philips monitor before, during (0 and 1 minute), and after the first outflow and inflow.
Oxygen Saturation Monitoring | 12 months
  Developed by the researchers, this form records oxygen saturation using a Philips monitor before, during (0 and 1 minute), and after the first outflow and inflow.
Parental Satisfaction | 12 months
  This researcher-developed questionnaire evaluates parent satisfaction with the non-pharmacological pain management method applied during the first inflow and outflow of PD. It consists of five yes/no questions. Each "yes" is scored as 1 and each "no" as 0, with total scores ranging from 0 to 10. Higher scores indicate greater satisfaction. The form will be completed after the first PD session

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Sağlık Bilimleri University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The data set will be shared online with other researchers during the data collection phase and while the data is being analyzed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months
Access Criteria: The third and fourth researchers will share data with the first and second researchers online during the data collection and analysis phases.
URL: https://camsakurasehir.saglik.gov.tr/TR-1111070/klinik-arastirmalar-etik-kurulu.html